CLINICAL TRIAL: NCT06280651
Title: Oral Health Implications of Dietary Preferences in Autistic Paediatric Population: A Cross-Sectional Study
Brief Title: Dietary Impacts on Oral Health in Autistic Children: A Cross-Sectional Analysis
Acronym: OHIDPAP-CS
Status: Not yet recruiting | Type: Observational
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, ASSITANT PROFESSOR, King Khalid University
Other Study IDs: RGP 2/348/44; RGP 2/348/44 (Other Grant/Funding Number: kING kHALID UNIVERSITY)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dental Caries in Children; Autistic Disorder; Dietary Habits
Keywords: Oral Health; Dietary Preferences; Autistic Paediatric Population; Oral Hygiene
MeSH Terms: conditions — Autistic Disorder; Feeding Behavior | interventions — Oral Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dietary preferences and their implications for oral health in children with Autism Spectrum Disorder — This study design typically does not involve interventions. Instead, it observes and analyzes existing conditions or behaviors-in this case, dietary preferences and their implications for oral health in children with Autism Spectrum Disorder (ASD)-without the researchers applying any specific treatment or experimental condition to the participants. The aim is to identify correlations or patterns at a specific point in time, rather than to assess the effects of an intervention.

SUMMARY:
The study aims to explore how dietary habits affect oral health in children with autism. By examining a cross-section of the autistic paediatric population, the research seeks to identify patterns or specific dietary preferences that may contribute to or mitigate oral health issues. This observational study does not intervene in participants' diets but observes existing habits and their oral health outcomes, aiming to provide insights that could guide better dietary recommendations and oral health practices for children with autism.

DETAILED DESCRIPTION:
The study investigates oral health implications of dietary preferences in autistic children, revealing diverse oral statuses and emphasizing tailored interventions. Key findings include significant associations between hygiene practices, periodontal disease, and dietary choices. The research highlights the need for personalized dental care, influenced by factors like age, gender, family income, parental education, and ASD severity. The study contributes to understanding oral health challenges in autistic children, suggesting dietary factors play a crucial role in oral health outcomes, calling for targeted strategies to improve their dental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 2 and 12 diagnosed with autism spectrum disorder are eligible to participate in the study.
* Informed consent from parents or legal guardians is a prerequisite.

Exclusion Criteria:

* Challenges that may impact study outcomes include coexisting medical conditions.
* Severe behavioral issues that may impede participation.
* Difficulties in obtaining informed consent, posing obstacles to comprehensive research endeavors.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study examines the impact of dietary habits on oral health among children with Autism Spectrum Disorder (ASD). It assesses how specific dietary choices correlate with oral health outcomes, including dental caries and periodontal disease. Key findings highlight the significance of diet in oral health management for autistic children, underscoring the need for specialized dietary advice and oral care strategies. The research aims to inform caregivers and healthcare professionals about the importance of monitoring and adjusting dietary habits to improve oral health in the ASD pediatric population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Assess the association between oral hygiene and periodontal disease severity to identify potential implications of dietary preferences for oral health status | 3 months
  This objective aims to explore how dietary habits among autistic pediatric populations influence oral health outcomes, particularly focusing on the correlation between oral hygiene practices and the severity of periodontal diseases. The study seeks to provide insights that could inform the development of targeted interventions and preventive strategies to address oral health issues in children with autism, emphasizing the impact of dietary choices on oral health.

IPD SHARING:
Plan to Share IPD: Undecided
The IPD Sharing Plan aims to advance research in oral health and dietary preferences in autistic children, ensuring data privacy. It includes sharing anonymized participant data (demographics, dietary habits, oral health status) and study methodologies. Data access requires a review for ethical soundness, a commitment to confidentiality, and is limited to affiliated researchers. This fosters collaboration while protecting participant information.